CLINICAL TRIAL: NCT05021653
Title: Exploration of the Role of Resilience and Its Development in Later Life Among HIV Infected Older Adults: a Qualitative Study
Brief Title: HIV Resilience Qualitative Study Hong Kong
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shui-Shan Lee, MD, Research Professor, Chinese University of Hong Kong
Other Study IDs: HKHIV resilience 01
Record Dates: First submitted 2021-08-16; First posted 2021-08-25 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: HIV Infections; Elderly Infection
Keywords: HIV; resilience; qualitative research; elderly
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men who have sex with men (MSM): Chinese men who have sex with men living with HIV infection and attending the service of HIV specialist service in Hong Kong
  Interventions: Other: no intervention
- non-MSM: Chinese heterosexual men and women living with HIV infection and attending the service of HIV specialist service in Hong Kong
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — No intervention involved

SUMMARY:
This qualitative study aims to explore lived experiences of older adults living with HIV in Hong Kong. Twenty older Chinese adults of age 50 or above will be recruited from an HIV specialist clinic providing HIV care in the public service. Qualitative, semi-structured interview will be conducted to explore risk factors contributing to life stress and adversity, and protective factors associated with resilience. The qualitative data will be delineated to propose a typology of older adults living with HIV as characterized by their unmet needs, barriers and facilitators of resilience-building.

DETAILED DESCRIPTION:
Objectives: The intersection of HIV and ageing has important implications for health and psychosocial wellbeing, which are complex in nature. In a setting with growing number of older adults living with HIV in Hong Kong, as in many other regions in the world, addressing their unmet healthcare needs is paramount. Failure to understand and recognise their needs will impede healthy ageing. This study aims to explore lived experiences of older adults living with HIV in regards their complex needs and resilience-building, with the specific objectives of examining associated factors of resilience development at individual-social- and structural level.

Design: A qualitative study targeting 20 older Chinese adults of age 50 or above who are living with HIV who are divided under the following groups: Group A: Chinese men who have sex with men and Group B: Chinese heterosexual males and females

Settings: Clinic providing HIV care in the public service

Methods: Participants will be recruited through purposive sampling based on their age (50-64; 65 and above of age), gender and sexual orientation. Qualitative, semi-structured interview will be conducted to explore: (1) risk factors contributing to life stress and adversity, and (2) protective factors associated with resilience. Interviews will be digitally recorded, transcribed verbatim and managed using "NVivo" software. Themes will be developed, constantly compared within and between targeted groups, using Grounded Theory approach.

Anticipated outcomes:

The qualitative data will be delineated to propose a typology of older adults living with HIV as characterized by their (1) unmet needs, (2) barriers of resilience-building, and (3) facilitators of resilience-building.

ELIGIBILITY:
Inclusion Criteria:

* Known and confirmed HIV infection
* age of 50 or above
* normally living in Hong Kong
* permanent residents of Hong Kong
* able to communicate in Cantonese

Exclusion Criteria:

* Active psychiatric disorder
* prisoners or under institutionalized care
* unable to give consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older adults living with HIV infection in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
risk items | 1 year
  risk factors contributing to stress and adversity
protective factors | 1 year
  Factors associated with resilience

CONTACTS AND LOCATIONS:
Overall Officials: Shui Shan Lee, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The descriptive data could only be accessed by the investigators and the research team, in line with the ethics approval obtained.